CLINICAL TRIAL: NCT06198699
Title: Effects of Jing Si Herbal Tea on Quality of Life and Sleep Among Patients With Dementia and Their Caregivers: A Randomized Controlled Trial
Brief Title: Effects of Jing Si Herbal Tea on Quality of Life and Sleep in Dementia and Their Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Collaborators: Buddhist Tzu Chi General Hospital (Other); Tzu Chi University (Other); E-DA Hospital (Other)
Responsible Party: Principal Investigator, Chung-Ying Lin, Associate Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCMF-JCT 113-03
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Dementia; Caregiver Burden; Quality of Life
Keywords: dementia; caregiver; quality of life; Jing Si Herbal Tea; psychosocial health; randomized controlled trial
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jing Si Herbal Tea Group (Experimental): Frequency: Two times of herbal tea (one in the morning; one in the afternoon) per day Duration: Consumption for three months Dosage: One pack (14g) with 600 ml water for each time of herbal tea consumption
  Interventions: Dietary Supplement: Jing Si Herbal Tea
- Barley Tea Group (Placebo Comparator): Frequency: Two times of barley tea (one in the morning; one in the afternoon) per day Duration: Consumption for three months Dosage: 600 ml each time of barley tea consumption
  Interventions: Dietary Supplement: Barley Tea

INTERVENTIONS:
Dietary Supplement: Jing Si Herbal Tea — Consuming Jing Si Herbal Tea for three months; twice per day with each time 14 g of Jing Si Herbal in 600 ml water
  Arms: Jing Si Herbal Tea Group
Dietary Supplement: Barley Tea — Consuming Barley Tea for three months; twice per day with each time 600 ml barley tea consumption
  Arms: Barley Tea Group

SUMMARY:
Jing Si Herbal Tea has been found to be effective in improving health for the conditions of cancers, aging, depression, and sleep. Such evidence has been shown in animal models and clinical research with publications in the international journals. However, empirical evidence regarding the effectiveness of Jing Si Herbal Tea for patients with dementia and their caregivers on their quality of life and psychosocial health remains unclear. Therefore, the present project aims to investigate the feasibility of taking Jing Si Herbal Tea among patients with dementia; then, to investigate if Jing Si Herbal Tea could improve quality of life and psychosocial health for patients with dementia and their caregivers. The project will be three years. The first year will examine the feasibility for the patients with dementia. A total of 100 patients with dementia will be recruited and they will be informed to take the Jing Si Herbal Tea two times per day (one time in the morning and another time in the afternoon). All the participants will be measured for their quality of life and psychosocial health at baseline, three months after baseline, and six months after baseline, to have initial evidence of the improvements in quality of life and psychosocial health without having a control group. The second year will recruit 200 patients with dementia and randomly assign them into a treatment group (taking Jing Si Herbal Tea) and a control group (taking placebo). All the participants will be measured for their quality of life and psychosocial health at baseline, three months after baseline, and six months after baseline, to investigate the strong evidence of Jing Si Herbal Tea on quality of life and psychosocial health. The third year will recruit 200 caregivers of patient with dementia and randomly assign them into a treatment group (taking Jing Si Herbal Tea) and a control group (taking placebo). All the participants will be measured for their quality of life and psychosocial health at baseline, three months after baseline, and six months after baseline, to investigate the strong evidence of Jing Si Herbal Tea on quality of life and psychosocial health.

ELIGIBILITY:
For people with dementia:

Inclusion Criteria:

* diagnosis of dementia
* 50 years or older
* with sufficient cognition to complete the questionnaires
* can communicate using Mandarin or Taiwanese

Exclusion Criteria:

* with renal function problems
* not suitable for Jing Si Herbal Tea after evaluation from a psychiatrist/physician
* with the condition of change the commencement of guardianship (or commencement of assistance)

For caregivers:

Inclusion Criteria:

* caregivers of people with dementia for more than half years
* 20 years or older
* with sufficient cognition to complete the questionnaires
* can communicate using Mandarin or Taiwanese

Exclusion Criteria:

* with renal function problems
* not suitable for Jing Si Herbal Tea after evaluation from a psychiatrist/physician
* with the condition of change the commencement of guardianship (or commencement of assistance)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Assessment for age (WHOQOL-AGE) [for people with dementia] | baseline; 3 months after baseline; 6 months after baseline
  quality of life measure; score range 13-65; higher score indicates better quality of life
Insomnia Severity Index [for both people with dementia and their caregivers] | baseline; 3 months after baseline; 6 months after baseline
  sleep problem measure; score range 0-28; higher score indicates more severe insomnia
World Health Organization Quality of Life Assessment brief version (WHOQOL-BREF) [for caregivers] | baseline; 3 months after baseline; 6 months after baseline
  quality of life measure; score range 4-20; higher score indicates better quality of life

SECONDARY OUTCOMES:
Katz Index of Independence in Activities of Daily Living [for people with dementia] | baseline; 3 months after baseline; 6 months after baseline
  activities of daily living function measure; score range 0-6; higher score indicates better activities of daily living
5 items of Geriatric Depression Scale [for people with dementia and their caregivers] | baseline; 3 months after baseline; 6 months after baseline
  depression measure; score range 0-5; higher score indicates greater depression
Short Portable Mental Status Questionnaire [for people with dementia] | baseline; 3 months after baseline; 6 months after baseline
  cognition measure; score range 0-10; higher score indicates poor cognition
Clinical Frailty Scale [for people with dementia] | baseline; 3 months after baseline; 6 months after baseline
  frailty measure; score range 1-9; higher score indicates more frail
Integrated care for older people [for people with dementia] | baseline; 3 months after baseline; 6 months after baseline
  intrinsic capacity measure; score range 0-13; higher score indicates poorer intrinsic capacity
Attitude and Thoughts Toward Older People Scale [for people with dementia and their caregivers] | baseline; 3 months after baseline; 6 months after baseline
  ageism measure; score range 17-85; higher score indicates higher level of ageism
Depression, Anxiety, Stress Scale-21 [for people with dementia and their caregivers] | baseline; 3 months after baseline; 6 months after baseline
  psychological distress measure; score range 0-63; higher score indicates greater distress
12 item of Zarit Burden Interview [for caregivers] | baseline; 3 months after baseline; 6 months after baseline
  caregiver burden measure; score range 0-48; higher score indicates greater burden

OTHER OUTCOMES:
Comorbidity | baseline
  Other chronic disease the participants have

IPD SHARING:
Plan to Share IPD: No